CLINICAL TRIAL: NCT01189058
Title: Modulation of Brain Plasticity After Perinatal Stroke: The PLASTIC CHAMPS Trial
Brief Title: Modulation of Brain Plasticity After Perinatal Stroke
Acronym: PLASTIC CHAMPS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Adam Kirton, Pediatric Neurologist, University of Calgary
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 22163
Record Dates: First submitted 2010-08-20; First posted 2010-08-26 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Stroke; Cerebral Palsy
Keywords: Perinatal stroke; Periventricular venous infarction; Presumed perinatal stroke; Neonatal stroke; Arterial ischemic stroke; Fetal stroke; Transcranial magnetic stimulation; Constraint-induced movement therapy; CIMT; Cerebral palsy; Congenital hemiplegia; Hemiplegic cerebral palsy; Neuroplasticity; Developmental plasticity
MeSH Terms: conditions — Stroke; Cerebral Palsy; Ischemic Stroke | interventions — Transcranial Magnetic Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rTMS and CIMT (Experimental): This group will receive both rTMS and CIMT.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS); Procedure: Constraint-induced movement therapy (CIMT)
- rTMS and no CIMT (Experimental): This group will receive rTMS only.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham and CIMT (Experimental): This group will receive CIMT and sham rTMS.
  Interventions: Procedure: Constraint-induced movement therapy (CIMT)
- Sham and no CIMT (No Intervention): This group will receive sham rTMS and no CIMT.

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS) — TMS can affect discrete functional ares of motor cortex offering non-invasive, painless mapping and modulation of motor systems. Inhibitory rTMS (1Hz)has been shown to safely lower motor cortex excitability in normal patients as well as adult and pediatric stroke patients. Dose is 20 minutes per day (1200 stimulations) x 10 days administered over the non-lesioned M1.
  Arms: rTMS and CIMT; rTMS and no CIMT
Procedure: Constraint-induced movement therapy (CIMT) — CIMT uses gentle restraint of the fully functional upper extremity to promote functional gains in the affected upper extremity. CIMT is well established to be safe and is likely effective in children with hemiplegic cerebral palsy, many of whom have perinatal stroke as studied here. A custom-fitted, bivalved cast is applied and worn for >90% of waking hours for the 2 weeks of active treatment according to protocol with daily assessments for comfort.
  Arms: Sham and CIMT; rTMS and CIMT

SUMMARY:
Newborn stroke is the leading cause of a common type of cerebral palsy (CP) that affects thousands of Canadian children and families. Treatments for CP are generally ineffective, and have traditionally focused on the weak body rather than the injured brain. Understanding how the newborn brain responds to injuries like stroke (plasticity) carries the greatest potential for better treatments. We propose to study the ability of two interventions to modulate brain plasticity toward better function in children with stroke-induced CP. One is a rehabilitation method called constraint-induced movement therapy (CIMT), the other is a type of non-invasive brain stimulation called transcranial magnetic stimulation (TMS). TMS is safe and comfortable for children and we recently showed it could improve motor function in children with stroke.

We will perform a special study to test both treatments simultaneously. Children 7-18 years with stroke-induced CP will be recruited into the study from across Alberta. Each child will randomly receive either TMS, CIMT, both, or neither each day for two weeks while attending our new HemiKids Power Camp for motor learning. Improvements will be measured by trained therapists over 1 year. TMS will also measure brain plasticity, both initially and following treatment. Our lead investigator is an expert in both newborn stroke and TMS and has assembled an experienced team of accomplished collaborators to ensure the completion of this important work. This will be the largest study of children with CP examined in this manner. This will be the first clinical trial of non-invasive brain stimulation (TMS) in CP, the largest trial of CIMT (and the first exclusive to newborn stroke), and the first study allowing the direct comparison of two different therapies. In establishing the first dedicated pediatric TMS laboratory in Canada, we will be the first to measure plasticity changes in newborn stroke, advancing new treatments of this previously untreatable and disabling disease.

Patient recruitment is currently underway at Alberta Children's Hospital. Application is currently underway to expand recruitment to Northern Alberta through the Glenrose Rehabilitation Hospital and Stollery Children's Hospital, to enable patients from Northern Alberta greater opportunity to participate as subjects in this study.

DETAILED DESCRIPTION:
Perinatal stroke is the leading cause of the most common term-born cerebral palsy: hemiplegic CP (HCP). With morbidity spanning all aspects of a child's life and lasting for decades, global impact is large. Mechanisms are poorly understood and prevention strategies remain elusive. Treatments are limited, leading to loss of hope in children and families that merits exploration of new interventions. Constraint-induced movement therapy (CIMT) may benefit but proper clinical trials are required. The investigators clinical-radiographic classifications have established perinatal stroke syndromes correlating with neurological outcome. Most common are: (1) arterial ischemic stroke of the middle cerebral artery (AIS-MCA) featuring cortical and subcortical damage acquired at birth and (2) periventricular venous infarction (PVI), a novel subcortical injury acquired in utero. These syndromes differ in the essential variables for plastic organization after perinatal injury: location and timing. In addition, recent animal and human studies suggest they may share a similar maladaptive plasticity whereby motor control of the weak side is "installed" in the non-lesioned hemisphere during development. Despite the ideal plasticity model such focal injury in a young brain provides, studies have been limited and suffer from small numbers of older patients with heterogeneous lesions. The value of studying plastic organization will be realized upon translation into meaningful patient benefits.

Transcranial magnetic stimulation (TMS) offers non-invasive measurement of the neurophysiological brain properties underlying neuroplasticity. Repetitive TMS (rTMS) may modulate such systems with therapeutic effect. the investigators recently demonstrated the ability of rTMS to improve motor function in children with chronic stroke. Advances in perinatal brain injury and neurodevelopment are, for the first time, affording novel windows of opportunity for interventions to direct plastic organization toward better outcomes. Via the Alberta Perinatal Stroke Project (APSP), the investigators propose a clinical trial of two interventions to improve function in HCP while measuring the fundamental neurophysiological properties at play.

Aim 1. Determine if rTMS and CIMT can improve motor function in HCP. Hypothesis: Two weeks of daily rTMS improves motor function at 30 days.

Aim 2. Define the neurophysiology of motor organization in stroke-induced HCP at baseline and following rTMS and CIMT.

Hypothesis: rTMS and CIMT reduce excitability of the non-lesioned motor cortex.

Population-based studies through the Alberta Perinatal Stroke Project (APSP) are establishing the largest perinatal stroke cohort to date. The investigators will complete a factorial 2 x 2 randomized clinical trial to determine the ability of daily rTMS and CIMT to improve motor function in children with HCP. Families will attend a child-centered, custom-designed intensive motor learning rehabilitation program (KidsCan Power Camp) for 2 weeks. Outcomes include validated measures of motor function and CP quality of life. The investigators will simultaneously measure the neurophysiology of plastic organization using TMS including cortical excitability, interhemispheric inhibition, and short interval intracortical inhibition. Baseline measures will define organization patterns while post-interventional measurement will evaluate the neurophysiological effects of rTMS and CIMT. Four groups of 16 children each (n=64) will be studied over 24 months with interim safety analysis after 10 and 32 patients.

Successful completion is assured by principle investigator experience in perinatal stroke and TMS and the collaborative support of world leaders in pediatric and adult stroke, TMS, basic neuroscience, and physiatry/rehabilitation. Understanding perinatal stroke plasticity and discovering methods to modulate it toward better outcomes carries a large impact, greatest for children with CP and their families.

ELIGIBILITY:
Inclusion criteria:

1. Symptomatic hemiplegic CP with impairment(s) of the upper extremity including the hand (Pediatric Stroke Outcome Measure motor >0.5; AND Manual Ability Classification System I, II,III, or IV; AND both child and parent perceive functional limitations (able to identify personally meaningful deficits in function).
2. MRI confirmed AIS-MCA or PVI (neuroradiological syndrome classified by two blinded, experienced investigators according to previously validated methods)
3. Age at enrollment: 6-18 years
4. Resident in province of Alberta for period of study
5. Informed consent/assent

Exclusion criteria:

1. Multifocal perinatal stroke or other brain injury/abnormality
2. Severe hemiparesis (no voluntary contraction in paretic hand, MACS level V)
3. Intellectual disability causing an inability to comply with study protocol
4. Unstable epilepsy (>1 seizure/month or >2 medication changes (dose or agent) in the last 6 months or history of recurrent status epilepticus)
5. Any TMS contraindication including implanted electronic devices
6. Botulinum toxin A injection in the affected upper extremity within the preceding 6 months
7. Orthopedic surgery in the affected upper extremity in the previous 12 months
8. Unwilling to delay any new therapeutic rehabilitational intervention directed towards upper limb function (aside from study home program) for the 6 month duration of the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM). | Completed 2 weeks or less before treatment day 1
  The COPM is an individualized, family-centered tool designed to guide participants to identify self-perception of difficulties in self-care, productivity (i.e school) and leisure activities.
Canadian Occupational Performance Measure (COPM) | Completed day 5 after treatment day 10
  The COPM is an individualized, family-centered tool designed to guide participants to identify self-perception of difficulties in self-care, productivity (i.e school) and leisure activities.
Canadian Occupational Performance Measure (COPM) | Completed 2 months after treatment day 10
  The COPM is an individualized, family-centered tool designed to guide participants to identify self-perception of difficulties in self-care, productivity (i.e school) and leisure activities.
Canadian Occupational Performance Measure (COPM) | Completed 6 months after treatment day 10
  The COPM is an individualized, family-centered tool designed to guide participants to identify self-perception of difficulties in self-care, productivity (i.e school) and leisure activities.

SECONDARY OUTCOMES:
PedsQL Cerebral Palsy Module version 3.0 Young child report (ages 5-7), Child report (ages 8-12), Teen report (ages 8-12) | Completed 2 weeks or less before treatment day 1
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health. The PedsQL-CP is a condition specific health related quality of life instrument validated for child self-report (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participants. The PedsQL-CP includes scales of: daily activities, school activities, movement/balance, pain/hurt, fatigue, eating activities, and speech/communication.
PedsQL Cerebral Palsy Module version 3.0 Young child report (ages 5-7), Child report (ages 8-12), Teen report (ages 8-12) | Completed 5 days after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health. The PedsQL-CP is a condition specific health related quality of life instrument validated for child self-report (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participants. The PedsQL-CP includes scales of: daily activities, school activities, movement/balance, pain/hurt, fatigue, eating activities, and speech/communication.
PedsQL Cerebral Palsy Module version 3.0 Young child report (ages 5-7), Child report (ages 8-12), Teen report (ages 8-12) | Completed 2 months after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health. The PedsQL-CP is a condition specific health related quality of life instrument validated for child self-report (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participants. The PedsQL-CP includes scales of: daily activities, school activities, movement/balance, pain/hurt, fatigue, eating activities, and speech/communication.
PedsQL Cerebral Palsy Module version 3.0 Young child report (ages 5-7), Child report (ages 8-12), Teen report (ages 8-12) | Completed 6 months after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health. The PedsQL-CP is a condition specific health related quality of life instrument validated for child self-report (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participants. The PedsQL-CP includes scales of: daily activities, school activities, movement/balance, pain/hurt, fatigue, eating activities, and speech/communication.
Pediatric Stroke Outcome Measure Short Neuro Exam Child Version (>2 years)(PSOM) | Completed before treatment day 1
  This is a validated outcome measure for perinatal and childhood stroke.
PedsQL Cerebral Palsy Module version 3.0 Parent Report for young child(ages 5-7), Parent Report for Child(ages 8-12), Parent report for teen(ages 8-12) | Completed 2 weeks or less before treatment day 1
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health from a parents perspective. The PedsQL-CP is a condition specific health related quality of life instrument validated for parent-report of their child (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participant's parents.
PedsQL Cerebral Palsy Module version 3.0 Parent Report for young child(ages 5-7), Parent Report for Child(ages 8-12), Parent report for teen(ages 8-12) | Completed day 5 after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health from a parents perspective. The PedsQL-CP is a condition specific health related quality of life instrument validated for parent-report of their child (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participant's parents.
PedsQL Cerebral Palsy Module version 3.0 Parent Report for young child(ages 5-7), Parent Report for Child(ages 8-12), Parent report for teen(ages 8-12) | Completed 2 months after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health from a parents perspective. The PedsQL-CP is a condition specific health related quality of life instrument validated for parent-report of their child (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participant's parents.
PedsQL Cerebral Palsy Module version 3.0 Parent Report for young child(ages 5-7), Parent Report for Child(ages 8-12), Parent report for teen(ages 8-12) | Completed 6 months after treatment day 10
  This instrument assesses domains of social/emotional well-being/acceptance, functioning, participation and physical health, access to services, pain and feelings about disability, and family health from a parents perspective. The PedsQL-CP is a condition specific health related quality of life instrument validated for parent-report of their child (5-18yrs). Version of PedsQL-CP used is age specific and will be completed by all participant's parents.
SHUEE (Shriners Hospital Upper Extremity Evaluation) | Completed 2 weeks or less prior to treatment day 1
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function in children with hemiplegic cerebral palsy. This tool includes spontaneous functional analysis and dynamic positional analysis and assesses the ability to perform grasp and release.
SHUEE (Shriners Hospital Upper Extremity Evaluation) | Completed day 5 after treatment day 10
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function in children with hemiplegic cerebral palsy. This tool includes spontaneous functional analysis and dynamic positional analysis and assesses the ability to perform grasp and release.
SHUEE (Shriners Hospital Upper Extremity Evaluation) | Completed 2 months after treatment day 10
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function in children with hemiplegic cerebral palsy. This tool includes spontaneous functional analysis and dynamic positional analysis and assesses the ability to perform grasp and release.
SHUEE (Shriners Hospital Upper Extremity Evaluation) | Completed 6 months after treatment day 10
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function in children with hemiplegic cerebral palsy. This tool includes spontaneous functional analysis and dynamic positional analysis and assesses the ability to perform grasp and release.
Box and Blocks Test | Completed 2 weeks or less before treatment day 1
  Tests the total number of blocks moved in 60 Seconds by each participant.
Box and Blocks Test | Completed 5 days after treatment day 10
  Tests the total number of blocks moved in 60 Seconds by each participant.
Box and Blocks Test | Completed 2 months after treatment day 10
  Tests the total number of blocks moved in 60 Seconds by each participant.
Box and Blocks Test | Completed 6 months after treatment day 10
  Tests the total number of blocks moved in 60 Seconds by each participant.
TMS Tolerability Measure | Completed 2 weeks or less before treatment day 1
  This child reportable tool evaluates potential side effects or unpleasant features a child may experience after receiving TMS or Sham. Children are also asked to rate their TMS or Sham experience using a 1(most pleasant or enjoyable)- 8(most unpleasant or unenjoyable) scale.
TMS Tolerability Measure | Completed 5days after treatment day 10
  This child reportable tool evaluates potential side effects or unpleasant features a child may experience after receiving TMS or Sham. Children are also asked to rate their TMS or Sham experience using a 1(most pleasant or enjoyable)- 8(most unpleasant or unenjoyable) scale.
TMS Tolerability Measure | Completed 2 months after treatment day 10
  This child reportable tool evaluates potential side effects or unpleasant features a child may experience after receiving TMS or Sham. Children are also asked to rate their TMS or Sham experience using a 1(most pleasant or enjoyable)- 8(most unpleasant or unenjoyable) scale.
TMS Tolerability Measure | Completed 6 months after treatment day 10
  This child reportable tool evaluates potential side effects or unpleasant features a child may experience after receiving TMS or Sham. Children are also asked to rate their TMS or Sham experience using a 1(most pleasant or enjoyable)- 8(most unpleasant or unenjoyable) scale.
Grip and Pinch Strength Measures (GS, PS) | Completed 2 weeks or less before treatment day 1
  Grip and pinch strength (GS, PS) are simple, quick measures of motor power, quantifiable with hand dynamometer that have been evaluated in children with Hemiplegic Cerebral Palsy.
Grip and Pinch Strength Measures (GS, PS) | Completed 5 days after treatment day 10
  Grip and pinch strength (GS, PS) are simple, quick measures of motor power, quantifiable with hand dynamometer that have been evaluated in children with Hemiplegic Cerebral Palsy.
Grip and Pinch Strength Measures (GS, PS) | Completed 2 months after treatment day 10
  Grip and pinch strength (GS, PS) are simple, quick measures of motor power, quantifiable with hand dynamometer that have been evaluated in children with Hemiplegic Cerebral Palsy.
Grip and Pinch Strength Measures (GS, PS) | Comopleted 6 months after treatment day 10
  Grip and pinch strength (GS, PS) are simple, quick measures of motor power, quantifiable with hand dynamometer that have been evaluated in children with Hemiplegic Cerebral Palsy.
Assisting Hand Assessment (AHA) | Completed 2 weeks or less before treatment day 1
  Assisting Hand Assessment (AHA) is a sensitive, reliable, and validated assessment of bi-manual tasks (functional assistive role of the weak hand) in children with HCP. The AHA has excellent clini-metric properties for evaluating bi-manual hand activities in HCP and pCIMT trials.
Assisting Hand Assessment (AHA) | Completed 5 days after treatment day 10
  Assisting Hand Assessment (AHA) is a sensitive, reliable, and validated assessment of bi-manual tasks (functional assistive role of the weak hand) in children with HCP. The AHA has excellent clini-metric properties for evaluating bi-manual hand activities in HCP and pCIMT trials.
Assisting Hand Assessment (AHA) | Completed 2 months after treatment day 10
  Assisting Hand Assessment (AHA) is a sensitive, reliable, and validated assessment of bi-manual tasks (functional assistive role of the weak hand) in children with HCP. The AHA has excellent clini-metric properties for evaluating bi-manual hand activities in HCP and pCIMT trials.
Assisting Hand Assessment (AHA) | Completed 6 months after treatment day 10
  Assisting Hand Assessment (AHA) is a sensitive, reliable, and validated assessment of bi-manual tasks (functional assistive role of the weak hand) in children with HCP. The AHA has excellent clini-metric properties for evaluating bi-manual hand activities in HCP and pCIMT trials.
Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) | Completed 2 weeks or less before treatment day 1
  A validated, criterion-referenced functional measure designed to detect therapeutic clinical change in children with HCP. Testing in children with moderate CP demonstrates high intra and inter-rater reliabilities and construct validity. We have demonstrated the utility of the MAUULF in the only previous rTMS trial in children 7-20 years with stroke-induced hemiparesis.
Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) | Completed 5 days after treatment day 10
  A validated, criterion-referenced functional measure designed to detect therapeutic clinical change in children with HCP. Testing in children with moderate CP demonstrates high intra and inter-rater reliabilities and construct validity. We have demonstrated the utility of the MAUULF in the only previous rTMS trial in children 7-20 years with stroke-induced hemiparesis.
Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) | Completed 2 months after treatment day 10
  A validated, criterion-referenced functional measure designed to detect therapeutic clinical change in children with HCP. Testing in children with moderate CP demonstrates high intra and inter-rater reliabilities and construct validity. We have demonstrated the utility of the MAUULF in the only previous rTMS trial in children 7-20 years with stroke-induced hemiparesis.
Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) | Completed 6 months after treatment day 10
  A validated, criterion-referenced functional measure designed to detect therapeutic clinical change in children with HCP. Testing in children with moderate CP demonstrates high intra and inter-rater reliabilities and construct validity. We have demonstrated the utility of the MAUULF in the only previous rTMS trial in children 7-20 years with stroke-induced hemiparesis.
ABILHAND-Kids -Manual ability measure | Completed 2 weeks or less before treatment day 1
  Measures manual ability in children (ages 6-15) with CP as perceived by the parents.
ABILHAND-Kids -Manual ability measure | Completed 5 days after treatment day 10
  Measures manual ability in children (ages 6-15) with CP as perceived by the parents.
ABILHAND-Kids -Manual ability measure | Completed 2 months after treatment day 10
  Measures manual ability in children (ages 6-15) with CP as perceived by the parents.
ABILHAND-Kids -Manual ability measure | Completed 6 months after treatment day 10
  Measures manual ability in children (ages 6-15) with CP as perceived by the parents.
The Revised Pediatric Motor Activity Log and the Tween Motor Activity Log (PMAL / TMAL) | Completed 2 weeks or less before treatment day 1
  Motor activity questionaire which asks parents to rate how often and how well their child uses his or her affected arm to complete some everyday activities. TMAL is used for Teenagers and PMAL is used for younger children.
The Revised Pediatric Motor Activity Log and the Tween Motor Activity Log (PMAL / TMAL) | Completed 5days after treatment day 10
  Motor activity questionaire which asks parents to rate how often and how well their child uses his or her affected arm to complete some everyday activities. TMAL is used for Teenagers and PMAL is used for younger children.
The Revised Pediatric Motor Activity Log and the Tween Motor Activity Log (PMAL / TMAL) | Completed 2 months after treatment day 10
  Motor activity questionaire which asks parents to rate how often and how well their child uses his or her affected arm to complete some everyday activities. TMAL is used for Teenagers and PMAL is used for younger children.
The Revised Pediatric Motor Activity Log and the Tween Motor Activity Log (PMAL / TMAL) | Completed 6 months after treatment day 10
  Motor activity questionaire which asks parents to rate how often and how well their child uses his or her affected arm to complete some everyday activities. TMAL is used for Teenagers and PMAL is used for younger children.
Biometrics Data Sheet | Completed each day during the 10 day camp program
  Records results of 3 groups of computer calibrated games 1. Eclipse which assesses pinch strength, 2. Space Shooter which assesses hand pronation and supination and 3. Balls and buckets which assesses wrist flexion and extension. Speed level, difficulty level, Range and percentage scores are recorded.
Paediatric Stroke Outcome Measure Short Neuro Exam (PSOM-SNE)-Child Version (Children Aged 2yrs and Older) | Completed before treatment day 1
  This neurological assessment tool assesses a child's: Level of Consciousness, Behaviour, Mental Status, Language, Cranial Nerves, Motor Movements, Tendon Reflexes, Fine Motor Coordination, Sensory and Gait, and rates any deficits using 0 (none), 0.5 (mild), 1.0 (Moderate) to 2 (severe) scale.
Home Program Log | Completed by each participant everyday during treatments days 1-10
  Participants are asked to complete a home log which records which activities, Part A (Functional goal areas with 2 hands for 10 minutes)and Part B (Strengthening activities with affected hand for 5 minutes) they have completed at home on a daily basis.
Home Program Log | Reassessed 2 months after treatment day 10
  Participants are asked to complete a home log which records which activities, Part A (Functional goal areas with 2 hands for 10 minutes)and Part B (Strengthening activities with affected hand for 5 minutes) they have completed at home on a daily basis.
Home Program Log | Reassessed 6 months after treatment day 10
  Participants are asked to complete a home log which records which activities, Part A (Functional goal areas with 2 hands for 10 minutes)and Part B (Strengthening activities with affected hand for 5 minutes) they have completed at home on a daily basis.
Camp Evaluation Form | Completed by participants on Day 10 of treatment
  This evaluation tool asked participants to rate their experience in attending the PLASTIC CHAMPS camp.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kirton, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Alberta Childrens Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Kirton A, Shroff M, Pontigon AM, deVeber G. Risk factors and presentations of periventricular venous infarction vs arterial presumed perinatal ischemic stroke. Arch Neurol. 2010 Jul;67(7):842-8. doi: 10.1001/archneurol.2010.140. PMID 20625091
- [Background] Kirton A, Deveber G, Gunraj C, Chen R. Cortical excitability and interhemispheric inhibition after subcortical pediatric stroke: plastic organization and effects of rTMS. Clin Neurophysiol. 2010 Nov;121(11):1922-9. doi: 10.1016/j.clinph.2010.04.021. PMID 20537584
- [Background] Kirton A, Wei X. Teaching neuroimages: confirmation of prenatal periventricular venous infarction with susceptibility-weighted MRI. Neurology. 2010 Mar 23;74(12):e48. doi: 10.1212/WNL.0b013e3181d5a47a. No abstract available. PMID 20308675
- [Background] Kirton A, deVeber G. Advances in perinatal ischemic stroke. Pediatr Neurol. 2009 Mar;40(3):205-14. doi: 10.1016/j.pediatrneurol.2008.09.018. PMID 19218034
- [Background] Kirton A, Chen R, Friefeld S, Gunraj C, Pontigon AM, Deveber G. Contralesional repetitive transcranial magnetic stimulation for chronic hemiparesis in subcortical paediatric stroke: a randomised trial. Lancet Neurol. 2008 Jun;7(6):507-13. doi: 10.1016/S1474-4422(08)70096-6. Epub 2008 May 1. PMID 18455961
- [Background] Kirton A, Deveber G, Pontigon AM, Macgregor D, Shroff M. Presumed perinatal ischemic stroke: vascular classification predicts outcomes. Ann Neurol. 2008 Apr;63(4):436-43. doi: 10.1002/ana.21334. PMID 18306227
- [Background] Kirton A, Westmacott R, deVeber G. Pediatric stroke: rehabilitation of focal injury in the developing brain. NeuroRehabilitation. 2007;22(5):371-82. PMID 18162700
- [Background] Raju TN, Nelson KB, Ferriero D, Lynch JK; NICHD-NINDS Perinatal Stroke Workshop Participants. Ischemic perinatal stroke: summary of a workshop sponsored by the National Institute of Child Health and Human Development and the National Institute of Neurological Disorders and Stroke. Pediatrics. 2007 Sep;120(3):609-16. doi: 10.1542/peds.2007-0336. PMID 17766535
- [Derived] Kirton A, Andersen J, Herrero M, Nettel-Aguirre A, Carsolio L, Damji O, Keess J, Mineyko A, Hodge J, Hill MD. Brain stimulation and constraint for perinatal stroke hemiparesis: The PLASTIC CHAMPS Trial. Neurology. 2016 May 3;86(18):1659-67. doi: 10.1212/WNL.0000000000002646. Epub 2016 Mar 30. PMID 27029628
- See also: Program Website — http://perinatalstroke.com/